CLINICAL TRIAL: NCT01137968
Title: A Randomized Phase II Study of Imetelstat as Maintenance Therapy After Initial Induction Chemotherapy for Advance Non-small Cell Lung Cancer(NSCLC)
Brief Title: Imetelstat as Maintenance Therapy After Initial Induction Chemotherapy in Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Geron Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP14B012
Record Dates: First submitted 2010-06-03; First posted 2010-06-07 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2015-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: imetelstat; imetelstat sodium; GRN163L; telomerase inhibitor; telomerase inhibition; maintenance therapy; non-small cell lung cancer; relapsed non-small cell lung cancer; advanced non-small cell lung cancer; NSCLC, cancer stem cells; Bevacizumab; post induction chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — imetelstat; GRN163L peptide; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- imetelstat plus standard of care (Experimental): imetelstat plus standard of care (bevacizumab or observation)
  Interventions: Drug: imetelstat; Drug: Bevacizumab
- Standard of care (Other): Bevacizumab or observation
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: imetelstat — 9.4 mg/kg over a 2 hour IV infusion on Day 1 and Day 8 of each 21 day cycle until disease progression.
  Other Names: GRN163L
  Arms: imetelstat plus standard of care
Drug: Bevacizumab — Dosage and duration will be according to the FDA-approved bevacizumab package insert. Bevacizumab will be administered on Day 1 of each 21-day cycle.
  Other Names: Avastin

SUMMARY:
The purpose of this is to evaluate the efficacy and safety of imetelstat (GRN163L) as maintenance therapy for patients with advanced stage NSCLC who have not progressed after 4 cycles of platinum based therapy.

Participants will be randomized in a 2:1 ratio to imetelstat + standard of care versus standard of care alone. Participants who received bevacizumab with their induction chemotherapy will continue to receive bevacizumab on this study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Ability and willingness to comply with requirements of the study protocol.
* Male or female, age 18 or over.
* Histologically or cytologically confirmed diagnosis of NSCLC
* Stage IV (using the 7th edition of AJCC, or wet IIIb / IV using the 6th edition), or recurrent locally advanced disease not amenable to radiation or surgery with curative intent and not amenable to concurrent chemoradiation.
* Patients have completed four to six cycles of platinum-based chemotherapy doublet for first line, advanced NSCLC, with no evidence of disease progression according to RECIST version 1.1. Adjuvant chemotherapy greater than one year prior to progression is allowed.
* Patients are willing and able to continue treatment with bevacizumab, if they received it with their platinum based chemotherapy.
* ECOG performance status 0-1
* Adequate bone marrow reserve as measured by ANC ≥ 1500/mm3, hemoglobin

  ≥ 9 g/dL, platelet count ≥ 75,000 μL. Must be measured ≥ 1 week after last transfusion of blood products and/or last dose of hematopoietic growth factor.
* Prothrombin time (PT) or INR or aPTT ≤ 1.5 x ULN.
* Serum creatinine < 1.5 mg/dL or creatinine clearance > 45 mL/min.
* Urinalysis with < 2+ protein or urinary excretion of < 2 g of protein/day (for patients to receive bevacizumab).
* AST (SGOT) and ALT (SGPT) < 2.5 x the ULN, (AST (SGOT) and ALT (SGPT) < 5 x the ULN if documented liver metastases).
* Serum bilirubin < 2.0 mg/dL (patients with Gilbert's syndrome: serum bilirubin < 3 x ULN).
* Alkaline phosphatase < 2.5 x ULN (patients with documented liver or bone metastases, alkaline phosphatase ≤ 5 x ULN).
* No other obvious related major organ toxicities which would compromise the patient's ability to participate in a clinical trial of a novel agent.
* Patients may have received prior radiation therapy for local or locally advanced disease providing that any clinically significant adverse effects associated with prior therapy have recovered to Grade 1 or less.
* Women of childbearing potential must have a negative serum pregnancy test and agree to use effective birth control during and for 12 weeks after the last treatment with imetelstat.
* Males must agree to use effective birth control for themselves or their partner during and for 12 weeks after the last treatment with imetelstat.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from screening and study entry:

* Patients who are not eligible for induction therapy with a platinum based chemotherapy doublet.
* Patients who have received, or are scheduled to receive pemetrexed or erlotinib as maintenance therapy.
* Patients receiving bevacizumab must not have a recent history of hemoptysis ≥ ½ teaspoon of red blood or history of ≥ 2 g/24 hr urine protein while receiving prior bevacizumab, or squamous cell histology.

Patients will be excluded from being randomized if any of the following criteria apply:

* Last dose of induction chemotherapy < 21 days prior to randomization or > 42 days prior to randomization
* History of pulmonary hemorrhage (> 1 teaspoon) within the 4 weeks prior to randomization.
* Anti-platelet therapy within 2 weeks prior to randomization, other than low dose aspirin prophylaxis therapy.
* Therapeutic anticoagulation therapy except for low dose warfarin (e.g., 1 mg by mouth per day).
* Radiation therapy within 3 weeks prior to randomization (palliative radiation therapy is allowed, provided that sites of bone marrow production, i.e. iliac crests are not in the radiation field)
* Major surgery within 4 weeks prior to first study drug administration (central line placement is allowed)
* Active central nervous system (CNS) metastatic disease. Patients with stable CNS disease following completion of radiation therapy and/or surgery are eligible.
* Any other active malignancy
* Active or chronically recurrent bleeding (e.g., active peptic ulcer disease)
* Clinically significant infection
* Active autoimmune disease requiring immunosuppressive therapy
* Clinically significant cardiovascular disease or condition including:
* Congestive heart failure (CHF) requiring therapy
* Need for anti-arrhythmic therapy for a ventricular arrhythmia
* Severe conduction disturbance
* Angina pectoris requiring therapy
* Medically uncontrolled hypertension per the Investigator's discretion
* Myocardial infarction within 6 months prior to first study drug administration
* New York Heart Association Class II, III, or IV cardiovascular disease
* Any other severe, acute, or chronic medical or psychiatric condition, laboratory abnormality, or difficulty complying with protocol requirements that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2010-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | From randomization to documented disease progression or death, whichever occurs earlier, through the end of the study period (8 mos. after the last participant is randomized)
  Defined as the time from randomization to documented disease progression or death, whichever occurs earlier,as determined by the Investigator's assessment according to RECIST, or death from any cause, whichever occurs earlier.

SECONDARY OUTCOMES:
Objective response | Occurring post randomization through end of study period (8 mos. after the last participant is randomized)
  Objective response (partial response plus complete response) occurring post-randomization as determined by the Investigator's assessment according to RECIST criteria using post-induction tumor dimensions as a baseline.
Time to all-cause mortality | From the date of randomization through end of study period (8 mos. after the last participant is randomized)
  Defined as the time from the date of radomization to death from any cause during the study period.
Safety and tolerability | From the date of randomization through the end of the study period (8 mos. after the last participant is randomized)
  Safety and tolerability will be assessed by the incidence, nature, and severity of adverse events, laboratory abnormalities, and vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Schiller, MD, Principal Investigator — University of Texas
Locations (33):
- United States (26):
  - Achieve Clinical Research, Llc, Birmingham, Alabama
  - Clearview Cancer Institute, Huntsville, Alabama
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - Cancer Care Associates of Fresno Medical Group Inc, Fresno, California
  - St. Joseph's Hospital, Orange, California
  - Kaiser Permanente Medical Center, Vallejo, California
  - University of Colorado Denver School of Medicine, Aurora, Colorado
  - Florida Cancer Specialists, Fort Myers, Florida
  - Integrated Community Oncology Network, Jacksonville, Florida
  - H. Moffitt Lee Cancer Center, Tampa, Florida
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Cancer Center of Kansas, Wichita, Kansas
  - Montgomery Cancer Center, Mount Sterling, Kentucky
  - Auerbach Hematology Oncology, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - Hematology Oncology Centers, Billings, Montana
  - Blumenthal Cancer Center, Charlotte, North Carolina
  - Kaiser Northwest, Portland, Oregon
  - South Carolina Oncology Associates, Columbia, South Carolina
  - The Jones Clinic, Germantown, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Scott and White Memorial Hospital (Texas A & M), Temple, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Northwest Medical Specialties, Tacoma, Washington
  - University of Wisconsin, Madison, Wisconsin
- Canada (2):
  - Hôpital Charles Lemoyne, Greenfield Park, Quebec
  - Hospital Notre-Dame, Montreal, Quebec
- Germany (5):
  - Krankenhaus Nordwest, Frankfurt, Frankfurt
  - Krankenhaus Grosshansdorf, Grosshansdorf, Hamburg
  - Universitaetsklinikum Mainz, Mainz, Mainz
  - Asklepios Klinik Gauting GmbH, Gauting, Munich
  - Klinikum rechts der Isar der TU München, München, Munich